CLINICAL TRIAL: NCT03743792
Title: The Effects of Acute Raspberry Intake on the Relationship Between Enhanced Metabolic Control and Cognitive and Psychomotor Function
Brief Title: Acute Raspberry Intake on Metabolic Control and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Human Nutrition Research Center on Aging (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 13165
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging; Age-related Cognitive Decline; Obesity
Keywords: Raspberry; Cognition; Vascular function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Freeze-dried red raspberry powder (25 g) in active breakfast meal
  Interventions: Dietary Supplement: Active breakfast
- Placebo (Placebo Comparator): Placebo breakfast
  Interventions: Dietary Supplement: Control breakfast

INTERVENTIONS:
Dietary Supplement: Active breakfast — freeze-dried red raspberry powder (12.5 g) in drink+ freeze-dried red raspberry powder (12.5 g) in buttermilk biscuit sandwich
  Arms: Active
Dietary Supplement: Control breakfast — Control drink + buttermilk biscuit sandwich
  Arms: Placebo

SUMMARY:
The purpose of this project is to determine whether restoring the post-prandial metabolic/inflammatory balance via supplementation with raspberries results in improved cognitive performance, and if these enhancements are mediated through improvements in vascular function.

DETAILED DESCRIPTION:
This study will investigate the effects of red raspberry in a relevant human model of metabolic disturbance to understand the relationship between red raspberry intake, metabolic and immune- balance and cognitive and psychomotor performance in older/over weight adults. A secondary goal of the project is to provide data on central vascular function in relation to metabolic-, inflammatory- and cognitive outcomes. Our primary working hypothesis is that red raspberries will improve metabolic- / inflammatory- balance in older overweight and obese adults resulting in improved cognitive and psychomotor performance mediated in part through improvements in vascular function. Two main objectives have been devised to meet the goals of the project and test our hypotheses: 1) Evaluate the effects of acute dietary raspberry intake on metabolic-associated impairments in cognitive and psychomotor function in overweight/obese adults (55-70y) following a meal challenge. 2) Evaluate the effects of acute dietary raspberry on measures of vascular function

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 35 kg/m2 and/or waist circumference (>35 inches for women, >40 inches for men)
* Aged 55-70 years old
* Able to provide informed consent and comply with study procedures
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial.
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.

Exclusion Criteria:

* Current smoker and/or marijuana user, past smokers may be allowed in the study if stopped >2 years
* Have a history or presence of atherosclerotic cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders
* Have recent surgery or injury to head
* Mini-Mental Status Exam score < 24 or Beck Depression Inventory score > 20
* Taking any medications that would interfere with outcomes of the study (i.e., lipid- lowering medications, anti-inflammatory drugs, and supplements, not including multivitamin/mineral or calcium/Vit D supplements),
* Unstable use of any medication/supplement
* Have a history of cancer in the prior 5 years, except for non-melanoma skin cancer
* Addicted to drugs and/or alcohol (>2 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Excessive exercisers or trained athletes
* Have allergies/intolerances to berries.
* Vegetarian/vegan or have extreme dietary habits.
* Excessive coffee/tea drinker
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Female who is pregnant, planning to be pregnant, breastfeeding
* Current regular consumption of berries which exceeds > 2 servings per day
* The individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Psychomotor function | Baseline to 6 hours
  Psychomotor function will be measured with the Grooved Pegboard

SECONDARY OUTCOMES:
Endothelial function | Baseline to 5 hours
  Vascular assessments will be measured using Near-infrared spectroscopy (NIRS)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Shukitt-Hale, PhD, Principal Investigator — USDA Human Nutrition Research Center on Aging; Tammy M Scott, PhD, Principal Investigator — Tufts University
Locations (1):
- USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No